CLINICAL TRIAL: NCT05571982
Title: Comparison of the Efficacy of Tidal Volume Breathing and Vital Capacity Breathing During High-flow Nasal Oxygen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2022-1017
Record Dates: First submitted 2022-10-06; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Adult Patients 20 Years of Age or Older Who Are Planning to Undergo Surgery Under General Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tidal volume breathing technique (Experimental): High-flow nasal oxygen will be applied to the patients through nasal openings using Optiflow system before anesthetic induction. Tidal volume breathing will be applied. Pulse oximetry, end-tidal O2, and oxygen reserve index will be monitored continuously.
  Interventions: Procedure: Tidal volume breathing technique
- Vital capacity breathing technique (Active Comparator): High-flow nasal oxygen will be applied to the patients through nasal openings using Optiflow system before anesthetic induction. Vital capacity breathing will be applied. Pulse oximetry, end-tidal O2, and oxygen reserve index will be monitored continuously.
  Interventions: Procedure: Vital capacity breathing technique

INTERVENTIONS:
Procedure: Tidal volume breathing technique — High-flow nasal oxygen will be applied to the patients through nasal openings using Optiflow system before anesthetic induction. Tidal volume breathing will be applied. Pulse oximetry, end-tidal O2, and oxygen reserve index will be monitored continuously.
  Arms: Tidal volume breathing technique
Procedure: Vital capacity breathing technique — High-flow nasal oxygen will be applied to the patients through nasal openings using Optiflow system before anesthetic induction. Vital capacity breathing will be applied. Pulse oximetry, end-tidal O2, and oxygen reserve index will be monitored continuously.
  Arms: Vital capacity breathing technique

SUMMARY:
The purpose of this study is to compare the preoxygenation efficacy of tidal volume breathing and vital capacity breathing.

ELIGIBILITY:
Inclusion Criteria:

-Adult patients 20 years of age or older who are planning to undergo surgery under general anesthesia

Exclusion Criteria:

-basal skull fracture, 2번 - facial anomaly, 3번 - consciousness disorder, 4번 - Risk of aspiration

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Oxygen reserve index | for 10 minutes before anesthetic induction. At Day 0.
  End-tidal O2 will be monitored continuously before anesthetic induction.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No